CLINICAL TRIAL: NCT01824550
Title: Exercise, Subclinical Atherosclerosis and Walking Mobility in Multiple Sclerosis
Brief Title: Home Exercise Intervention in Persons With Multiple Sclerosis
Acronym: HOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Bo Fernhall, Dean and Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-0836; RG 4702A1/2 (Other Grant/Funding Number: NMSS)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- home-based exercise training condition (Experimental): Home based endurance exercise training
  Interventions: Other: home-based exercise training condition
- attention control condition (No Intervention): Attention control condition - home based flexibility training

INTERVENTIONS:
Other: home-based exercise training condition — Home based endurance exercise training
  Arms: home-based exercise training condition

SUMMARY:
The objective of this study is to determine the effect of home-based, aerobic exercise training on subclinical atherosclerosis and mobility disability in persons with Multiple Sclerosis (MS). Our central hypothesis is that aerobic exercise training reduces both subclinical atherosclerosis and mobility disability.

DETAILED DESCRIPTION:
This study will use a two-arm randomized control trial (RCT) design to examine the effect of a home-based exercise training program versus a minimal exercise, attention control condition on markers of subclinical atherosclerosis and mobility disability in persons with MS. The primary outcomes will be subclinical atherosclerosis including measures of arterial structure and function and measures of mobility disability including the six-minute walk and timed 25-foot walk, GaitRite walking assessment and one week of accelerometry data.

Fifty-four persons with MS who have an Expanded Disability Status Score (EDSS) score between 0 and 4.0 will be randomized into either the home-based exercise training condition or the attention control condition. Participation in this study will include a 3-month exercise program to be completed at home. In addition, participants will need to come to University of Illinois at Chicago (UIC) three times to undergo testing. Each visit will take about 3-4 hours to complete. Testing that will take place during these three visits include blood pressure measurement, six vascular (artery) measurements, heart measurements, short walking tests, peak aerobic capacity test, blood draw, five quality of Life questionnaires and two cognitive function tests.

The home-based exercise regimen will include cycle ergometry as an aerobic mode of training 3 times per week with a gradual progression of duration and intensity across a 12-week period. Exercise prescription will be based on the peak aerobic capacity cycling test conducted during the first visit. The attention control will involve stretching using the same frequency and duration across a 12-week period with exercises recommended by the National Multiple Sclerosis Society (NMSS). Both arms will receive weekly internet "coaching" sessions via video chatting.

Subclinical atherosclerosis and mobility disability data will be collected before, after 6 weeks of training and immediately after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* physically inactive
* BMI<40
* 1st stage of MS (i.e., defined as EDSS score of 0 - 4.0)
* independently ambulatory (walking without an assistive device such as a cane or orthotic)
* relapse free in the past 30 days
* confirmed diagnosis of MS
* asymptomatic (i.e., no underlying clinically diagnosed cardiovascular disease)
* be on a stable disease modifying therapy
* physician approval for undertaking exercise testing and training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Subclinical atherosclerosis | 3 months
  This will me measured through carotid intima media thickness, flow mediated dilation of forearm, and aortic pulse wave velocity

SECONDARY OUTCOMES:
Mobility disability | 3 months
  This will be measured by the 6-min walk, 25 ft walk, the "Get-up-and-go" test and by gait characteristics.

OTHER OUTCOMES:
Disease state, and fatigue | 3 months
  This will be measured via questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fernhall, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States